CLINICAL TRIAL: NCT03157583
Title: Determination of the Sun Protection Factor (SPF) and in Vitro UVA Protection Factor (UVAPF) of Four Developmental Sunscreen Formulations
Brief Title: A Study to Measure the Sun Protection Factor (SPF) and Ultraviolet-A Protection Factor (UVAPF) of Four Developmental Sunscreen Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207583
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-05

CONDITIONS: Sunscreening Agents
MeSH Terms: interventions — Glycerol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Reference product (for SPFi calculation) (Active Comparator): This arm will include all the test sites on the participants back where reference product (P3 standard sunscreen) will be applied.
  Interventions: Other: P3 Standard, (Expected SPF 16)
- Test product 1 (Experimental): This arm will include all the test plates used for UVAPF testing and test sites on the participants back where test product 1 will be applied for SPF testing.
  Interventions: Other: NGBUV000A, (Expected SPF 30)
- Test product 2 (Experimental): This arm will include all the test plates used for UVAPF testing and test sites on the participants back where test product 2 will be applied for SPF testing.
  Interventions: Other: NGBUV000B, (Expected SPF 30)
- Test product 3 (Experimental): This arm will include all the test plates used for UVAPF testing and test sites on the participants back where test product 3 will be applied for SPF testing.
  Interventions: Other: NGBUV000C, (Expected SPF 30)
- Test product 4 (Experimental): This arm will include all the test plates used for UVAPF testing and test sites on the participants back where test product 4 will be applied for SPF testing.
  Interventions: Other: NGBUV000D, (Expected SPF 30)
- Negative control (for SPFi calculation) (No Intervention): This arm will include all the test sites on the participants back which will be left unprotected.
- Reference (for UVAPFi calculation) (Active Comparator): This arm will include test plates treated with reference sunscreen formulation S2.
  Interventions: Other: Sunscreen formulation S2
- Blank control (for UVAPFi calculation) (Other): This arm will include blank test plates treated with glycerin.
  Interventions: Other: Glycerin

INTERVENTIONS:
Other: NGBUV000A, (Expected SPF 30) — A total of 2.0 ± 0.05 mg/cm2 (milligram per centimeter square of test site area) NGBUV000A (test product 1) will be spread at the topical test sites on the back of each participant. And a total of 1.3 mg/cm2 of test product 1 will be applied to the test plates.
  Arms: Test product 1
Other: NGBUV000B, (Expected SPF 30) — A total of 2.0 ± 0.05 mg/cm2 NGBUV000B (test product 2) will be spread at the topical test sites on the back of each participant. And a total of 1.3 mg/cm2 of test product 2 will be applied to the test plates.
  Arms: Test product 2
Other: NGBUV000C, (Expected SPF 30) — A total of 2.0 ± 0.05 mg/cm2 NGBUV000C (test product 3) will be spread at the topical test sites on the back of each participant. And a total of 1.3 mg/cm2 of test product 3 will be applied to the test plates.
  Arms: Test product 3
Other: NGBUV000D, (Expected SPF 30) — A total of 2.0 ± 0.05 mg/cm2 NGBUV000D (test product 4) will be spread at the topical test sites on the back of each participant. And a total of 1.3 mg/cm2 of test product 4 will be applied to the test plates.
  Arms: Test product 4
Other: P3 Standard, (Expected SPF 16) — A total of 2.0 ± 0.05 mg/cm2 reference P3 standard will be spread at the topical test sites on the back of each participant.
  Arms: Reference product (for SPFi calculation)
Other: Sunscreen formulation S2 — A total of 1.3 mg/cm2 of sunscreen formulation S2 will be applied to the test plates.
  Arms: Reference (for UVAPFi calculation)
Other: Glycerin — A total of 1.3 mg/cm2 of glycerin will be applied to the test plates.
  Arms: Blank control (for UVAPFi calculation)

SUMMARY:
The purpose of this study is to determine the SPF and UVAPF of four sunscreen formulations using international standard methodologies ISO24444:2010 for SPF and ISO24443:2012 for UVAPF.

DETAILED DESCRIPTION:
This study consist of two steps. Step 1: determination of the SPF of the test products which will be performed as a single-center, randomized, evaluator blind, intra-individual comparison, no treatment and positive controlled clinical study as per ISO24444:2010. And Step 2: determination of the UVAPF of the test products which will be performed as a single center, open-label, negative and positive controlled technical test as per ISO24443:2012 (using test plates for assessing UV transmittance of four developmental sunscreens).

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical examination
* Participants with a Fitzpatrick Skin Type of I, II or III
* Participants with an Individual Typology Angle (ITA°) greater than 28°

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding or lactating
* Participants having used medication with known photo-toxic and/or photosensitizing potential (e.g. hypericum perforatum, antibiotics, blood pressure regulating agents) up to 14 days prior to screening
* Participants with a history of systemic therapy with anti-inflammatory agents or analgesics (e.g. diclofenac) up to 3 days prior to screening
* Participants with dermatological conditions
* Participants with a history of abnormal response to the sun
* Participants having marks, blemishes or nevi or presenting existing sun damage in the test area
* Participants having excessive hair, moles, tattoos, scars or other imperfections in the test area that could influence the investigation
* Participants with a history of systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines (e.g. anti-allergics) up to 7 days prior to screening
* Participants with a non-uniform skin colour or hyperpigmentation in the test area
* Participants with a medical history of dysplastic nevi or melanoma
* Participants with one of the following illnesses that might require regular systemic medication: Insulin-dependent diabetes, cancer
* Participants with asthma, unless medicated
* Participants with an electronic implant (e.g. pace maker, insulin pump, hearing aid) that cannot be removed during irradiation
* AIDS (acquired immune deficiency syndrome) and infectious hepatitis, if known to the participants
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Known allergy to latex
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days prior to screening
* Participation in another clinical study involving UV exposure to the same test site up to 2 months prior to screening
* Previous participation in this study
* Recent history (within the last 5 years) of alcohol or other substance abuse
* Participants who have used a tanning bed or other tanning treatment on the back area up to 1 month prior to screening
* Participants accustomed to using tanning beds
* Participants who have used self-tanning products on the back area in the previous 1 month prior to screening
* An employee of the sponsor or the study site or members of their immediate family

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Schenefeld, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were enrolled at one center in Germany.
Pre-assignment Details: Total of 9 participants were screened for the study out of which 1 participant did not meet the study criteria. Remaining 8 participants were randomized in the study.
Groups:
- All Participants: All the participants randomized to the study. In this study, there were a total of 7 test sites assigned to each participant. One test site was used for provisional MEDu (Minimal Erythemal Dose of Unprotected Skin) measurement, on the remaining 6 sites test products (4) and the positive control product (P3 standard) were applied and 1 site was left unprotected.
Period: Overall Study
Arm/Group | All Participants
Started | 8
Completed | 7
Not Completed | 1
Not completed — Other (did not meet study criteria) | 1

BASELINE CHARACTERISTICS:
Population: Baseline parameters were reported for safety population (N=8). The Safety population included all participants who applied any of the study products.
Groups:
- All Participants: Included all the participants who randomized to receive the study product.
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (18.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Arithmetic Mean of Individual Sun Protection Factor (SPFi) Values
Description: Arithmetic mean of all valid SPFi values of each product on each participant was calculated from the individual Minimal Erythemal Dose (MED) on product treated (MEDp) test sites in relation to unprotected (MEDu) test sites 16-24 hours after exposure to ultraviolet (UV) radiation. SPFi = MEDp/MEDu. No inferential statistical analysis was performed for this outcome.The provisional MEDu was the lowest dose of UV radiation that produces the first perceptible unambiguous erythema with defined borders appearing over most of the field of UV exposure.Higher values represents increased SPF protection.
Time Frame: Up to 24 hours post UV exposure
Population: Analysis population included all randomized participants who underwent irradiation at Visit 4. Here, number analyzed signifies participants with available data for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: Ratio
Groups:
- Test Product 1: This arm included all the test sites on the participants back where test product 1 was applied for SPF testing.
- Test Product 2: This arm included all the test sites on the participants back where test product 2 was applied for SPF testing.
- Test Product 3: This arm included all the test sites on the participants back where test product 3 was applied for SPF testing.
- Test Product 4: This arm included all the test sites on the participants back where test product 4 was applied for SPF testing.
- Reference Product (for SPFi Calculation): This arm included all the test sites on the participants back where reference product (P3 standard sunscreen) was applied.
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4 | Reference Product (for SPFi Calculation)
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
Ratio | 33.1 [26.08 to 40.22] | 35.2 [25.85 to 44.42] | 35.2 [26.82 to 43.68] | 45.2 [38.80 to 51.58] | 15.6 [12.66 to 18.59]

2. Secondary Outcome: Spectrum of Sun Protection
Description: Broad spectrum of sun protection was calculated by the ratio of the arithmetic mean of SPF to the arithmetic mean of UVAPF. Higher values represents increased SPF protection.
Time Frame: Up to 30 minutes post UV exposure
Population: Analysis population included all randomized participants who underwent irradiation at Visit 4.
Measure: Number; unit: Ratio
Groups:
- Test Product 1: This arm included all the test plates used for UVAPF testing and test sites on the participants back where test product 1 was applied for SPF testing.
- Test Product 2: This arm included all the test plates used for UVAPF testing and test sites on the participants back where test product 2 was applied for SPF testing.
- Test Product 3: This arm included all the test plates used for UVAPF testing and test sites on the participants back where test product 3 was applied for SPF testing.
- Test Product 4: This arm included all the test plates used for UVAPF testing and test sites on the participants back where test product 4 was applied for SPF testing.
- Reference (for UVAPFi and SPFi Calculation): This arm included test plates treated with reference sunscreen formulation S2. Also includes all the test sites on the participants back where reference product (P3 standard sunscreen) was applied.
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4 | Reference (for UVAPFi and SPFi Calculation)
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
Ratio | 3.11 | 2.98 | 2.88 | 2.95 | 1.13

ADVERSE EVENTS:
Time Frame: Approximately 16 days
Groups:
- Negative Control (for SPFi Calculation): This arm included all the test sites on the participants back which were left unprotected.
Arm/Group | Reference Product (for SPFi Calculation) | Negative Control (for SPFi Calculation) | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT03157583/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT03157583/SAP_001.pdf